CLINICAL TRIAL: NCT07097857
Title: Assessment of Revascularization in Plantar Foot of Diabetic Mellitus Patients Pre and Post Angioplasty Using Spatial Frequency Domain Imaging
Brief Title: Assessment of Revascularization in Plantar Foot of Diabetic Patients Pre and Post Angioplasty Using Spatial Frequency Domain Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/2648
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Arterial Disease(PAD); Imaging Evaluation
Keywords: Spatial Frequency Domain Imaging; Peripheral Arterial Disease; Non-invasive imaging
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Spatial Frequency Domain Imaging (SFDI) Imaging pre and post-ll angioplasty
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SFDI Imaging (Experimental): SFDI Imaging performed on both ipsilateral and contralateral foot. Imaging repeated on heel and pad regions of foot.
  Interventions: Other: SFDI

INTERVENTIONS:
Other: SFDI — SFDI imaging is performed on both treated and untreated limb.

SUMMARY:
To explore the usefulness of SFDI in the assessment of revascularization pre and post intervention

DETAILED DESCRIPTION:
Diabetes is a chronic disease with high cardiovascular morbidity and mortality ((Matheus et al., 2013)). Approximately 150 million worldwide are suffering from this condition and the number is expected to rise to 300 million by 2025. In Singapore, diabetes is the 10th leading cause of death accounting for 1.7 per cent total deaths in 2011. By 2030, the number of Singapore residents above 40 with diabetes is projected to increase by another 200,000 from about 400,000 today (Diabetes in Singapore: Stats and Prevention Tips - HealthXchange, n.d.). Despite having one of the world's highest life expectancies and a modern health care system, Singapore has one of the highest rates of lower extremity amputation (LEA) in the world, with public hospitals here needing to conduct some four amputation procedures a day ((Amputation of Limbs Regarded as a Last Resort - Singapore General Hospital, n.d.)).

However, patients who seek treatment early enough have the option of various intervention treatments to salvage limbs. These include re-vascularisation (angioplasty or bypass) and treatment of infection (drainage of abscesses or debridement). In Singapore, limb salvage therapies have led to a 20% reduction in LEA operations in 2015 compared to the year before ((SINGAPORE: ONE OF WORLD'S HIGHEST FOR DIABETES-RELATED LEG AMPUTATIONS, n.d.)). Unfortunately, the clinical success of these procedures in diabetics drop to 69% at 12 months (Lazaris et al., 2004). This is owing to the lack of objective feedback of limb perfusion. Non invasive imaging modalities that predict outcomes of such revascularization procedures can help in early intervention and thus limb salvage. Recently, SFDI, a noninvasive optical imaging method capable of measuring tissue oxygen saturation (StO2) and tissue haemoglobin has been show to predict diabetic foot ulcer onset in the US population (Lee et al., 2020). Herein, we hypothesize that these microvasculature information offered by SFDI can be used to predict the outcomes of revascularization procedures. To test this hypothesis, we propose an exploratory pilot study to use SFDI on 15 diabetic patients undergoing lower limb revascularization and acquire images of the plantar foot before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 21 years and above with diabetes and undergoing lower limb arterial angioplasty
* Willingness to participate in the study and undergo foot physiological assessments using SFDI

Exclusion Criteria:

* Mentally incompetent, younger than 21 years of age, prisoners, pregnant or breastfeeding women
* Patients unable to provide informed consent
* Any medical condition which makes the candidate an inappropriate subject for study participation, in the investigator's judgment

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in perfusion measured by tissue oxygen saturation | Pre and Post angioplasty on Day 0
  Change in perfusion is assessed by level of tissue oxygen saturation measured pre and post revascularization to evaluate the usefulness of SFDI in the assessment of revascularization pre and post intervention.

SECONDARY OUTCOMES:
Compare SFDI measurements to Toe Pressure | Pre and Post angioplasty on Day 0
  Toe Pressure measurements are done pre and post-op and compared against SFDI values obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Tze Tec Chong, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, SG, Singapore

IPD SHARING:
Plan to Share IPD: No
All data is protected by Personal Data Protection Act.

REFERENCES:
- [Background] Lee S, Mey L, Szymanska AF, Takhar HS, Cuccia DJ, Mazhar A, Yu K. SFDI biomarkers provide a quantitative ulcer risk metric and can be used to predict diabetic foot ulcer onset. J Diabetes Complications. 2020 Sep;34(9):107624. doi: 10.1016/j.jdiacomp.2020.107624. Epub 2020 May 19. PMID 32522482
- [Background] Amputation of limbs regarded as a last resort - Singapore General Hospital. (n.d.). Retrieved June 29, 2021, from https://www.sgh.com.sg/news/patient-care/amputation-of-limbs-regarded-as-a-last-resort